CLINICAL TRIAL: NCT05062954
Title: Effects of a Polyphenol-rich Cranberry Extract on Cardiometabolic and Neurocognitive Health in Individuals With Abdominal Obesity: a Double-blind Randomized Controlled Trial
Brief Title: Effects of a Polyphenol-rich Cranberry Extract on Cardiometabolic and Neurocognitive Health
Acronym: Neurocan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 128976
Record Dates: First submitted 2021-08-31; First posted 2021-09-30 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Abdominal Obesity
MeSH Terms: conditions — Obesity, Abdominal | interventions — Proanthocyanidins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Polyphenol-rich cranberry extract supplement standardized in PACs (Experimental): Supplementation with polyphenol-rich cranberry extract standardized in PACs (1 capsule / day)
  Interventions: Dietary Supplement: Polyphenol-rich cranberry extract supplement standardized in proanthocyanidins
- Placebo supplement (Placebo Comparator): Supplementation with placebo (1 capsule / day)
  Interventions: Dietary Supplement: Placebo supplement

INTERVENTIONS:
Dietary Supplement: Polyphenol-rich cranberry extract supplement standardized in proanthocyanidins — Participants will be randomly assigned to the consumption of one capsule of Polyphenol-rich cranberry extract standardized in PACs.
  Arms: Polyphenol-rich cranberry extract supplement standardized in PACs
Dietary Supplement: Placebo supplement — Participants will be randomly assigned to the consumption of one capsule of placebo per day for 56 consecutive days.
  Arms: Placebo supplement

SUMMARY:
The objective of this double-blind, parallel, randomized placebo-controlled clinical trial is to evaluate the effects of consumption of polyphenol-rich cranberry extract standardized in PACs (36 mg PACs/capsule) on cardiometabolic and neurocognitive health in women and men presenting abdominal obesity over an 8-week intervention period.

The study will be conducted at Quebec Heart and Lung Institute - Laval University. The study will involve a total of 60 adult men and women presenting abdominal obesity. Included participants will be randomly assigned to the consumption of a cranberry extract or a placebo at a rate of one capsule per day for 8 weeks (56 days). The main outcomes are changes in metabolic profile, neurocognitive performance as well as brain structure and function following polyphenol-rich cranberry extract standardized in PACs compared with the placebo.

DETAILED DESCRIPTION:
Background :

Abdominal obesity is associated with impaired cognitive function and increased risk of neurodegenerative diseases. The metabolic disorders associated with obesity may lead to alterations in brain function and structure, explaining the link between obesity and some cognitive dysfunction. Magnetic resonance imaging (MRI) studies show that obese individuals are characterized by gray matter atrophy in brain regions involved in self-control. Atrophy and alteration of white matter fibers have also been observed in these individuals. However, the mechanisms explaining these changes are not yet elucidated. It has been suggested that metabolic and inflammatory alterations associated with abdominal obesity may lead to these brain alterations.

It is well known that dietary intake influences the composition and diversity of the gut microbiota and that its disruption plays a central role in the development of obesity, chronic low-grade inflammation, insulin resistance and cardiovascular disease. Some studies have reported improvements in blood pressure, lipid profile, glucose homeostasis, endothelial function, arterial stiffness and inflammation following cranberry consumption, but others found no significant changes. A recent meta-analysis reported that taking a polyphenol-rich supplement is associated with improved cognitive function in young adults. Although the mechanisms underlying the beneficial effects of polyphenols on brain function and cognition remain to be elucidated, some studies suggest that these effects may be associated with their anti-inflammatory and antioxidant properties and their possible effect on the cerebrovascular system. To our knowledge, there are no randomized controlled studies that have evaluated the effects of polyphenol-rich cranberry extract standardized in PACs on neurometabolic and neurocognitive functions in participants with abdominal obesity.

Objectives and Hypothesis:

The objective of this double-blind, randomized placebo-controlled clinical trial is to evaluate the effects of consumption of polyphenol-rich cranberry extract standardized in PACs (36 mg PACs/capsule) on cardiometabolic and neurocognitive health in abdominally obese women and men over an 8-week period.

The overall hypothesis is that standardized extract of PACs from cranberry improves the metabolic profiles in abdominally obese individuals and this will have a beneficial impact on brain and neurocognitive functions.

Methodology:

Sixty men and women with a BMI equal or greater than 25 kg/m2 and an altered blood lipid profile (triglycerides) will be recruited at the IUCPQ-Université Laval via social networks and Laval University's recall lists. The study will include 3 visits to the IUCPQ-Université Laval as well as the consumption of a cranberry extract or a placebo at a rate of one capsule per day for 8 weeks (56 days). The eligibility visit (V1) consists of completing a medical history questionnaire, and anthropometric and fasting blood lipid measurements. Individuals eligible to participate will then be invited to 2 identical visits at the IUCPQ-Université Laval (V2 and V3). At visit 2, cognitive tasks, anthropometric measurements, blood pressure, MRI (Philips 3T) and a pan-body DXA will be performed in all participants. Cognitive function will be measured using a battery of validated neurocognitive tasks. On the morning of each MRI session, fasting blood samples will be collected. Stool samples will be collected by participants prior to each visit 2 and 3 to measure microbiota composition. Following visit 2, participants will leave with capsules of cranberry extract containing 36 mg of PACS or a placebo (double-blind randomization) and will be asked to consume one capsule per day for 56 consecutive days. They will return for the 3rd visit (identical to V2) 8 weeks after starting the supplements. Dietary and physical activity questionnaires will also be completed online before visits 2 and 3. At the beginning of the visits, any changes in the participant's health condition and use of medications and natural health products will be documented. A follow-up phone call will be scheduled with each participant on day 28 of the intervention to ensure that the intervention is going well. Adverse events related to supplementation will be documented. An end-of-study questionnaire will be completed by the participant at the last visit (V3) to confirm study blinding. Participants will be asked to report the remaining capsules at the last visit (V3), which will allow assessment of compliance with the intervention.

ELIGIBILITY:
Inclusion criteria:

* Men and women aged between 30-70 years old;
* BMI equal or greater than 25 kg/m2;
* Waist circumference ≥85 cm for women, ≥90 cm for men;
* Stable weight in the past 3 months;
* Plasma triglycerides levels ≥1.5 mmol/L for men and women;
* Access to a computer and Internet.

Exclusion criteria:

* Any severe uncontrolled medical, surgical, neurological or psychiatric condition;
* Medication for dyslipidemias, CVD, T2D or obesity;
* Medication that may affect the CNS;
* Gastro-intestinal conditions or disorders likely to impact on absorption;
* History of nephrolithiasis or urolithiasis;
* Contraindications to MRI (cardiac pacemaker/defibrillator, cochlear implant or other ear implant, implanted insulin pump or other infusion pump systems, neurostimulator or other electronic/magnetic implant or device, any type of prothesis, aneurysm clips, any metallic fragments, vascular access port, catheter, dental retainer, claustrophobia, surgery in the last 3 months);
* Anticoagulant/blood thinning medication in the last month;
* Pregnant or breastfeeding women;
* Substance or alcohol abuse;
* Known allergy or intolerance to cranberry;
* Currently smoking.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-21 (Actual); Primary Completion 2023-08 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Changes in basic plasma lipid-lipoprotein profile | 8 weeks
  Fasting blood samples
Changes in glucose homeostasis | 8 weeks
  Fasting blood samples
Changes in lipopolysaccharide binding protein (LBP) | 8 weeks
  Fasting blood samples
Changes in white matter health assessment | 8 weeks
  T2-weighted images, axial fluid-attenuated inversion recovery
Changes in brain density in key regions | 8 weeks
  Structural MRI measurements
Changes in functional brain connectivity | 8 weeks
  Resting state functional MRI
Changes in white matter integrity | 8 weeks
  Diffusion tensor imaging
Changes in cerebral vasculature | 8 weeks
  Magnetic resonance angiography time-of-flight (MRA-TOF)
Gut microbiota composition | 8 weeks
  Measures in fecal samples

SECONDARY OUTCOMES:
Changes in executive function | 8 weeks
  Stroop
Changes in attention span and short-term working memory | 8 weeks
  Digit Span
Changes in cognitive flexibility and speed of information processing | 8 weeks
  Trail Making Test (Parts A and B)
Changes in biomarkers of gut endotoxemia | 8 weeks
  Blood plasma samples will be analysed for presence of lipopolysaccharide (LPS)
Changes in biomarkers of gut permability | 8 weeks
  Blood plasma samples will be analysed for presence of zonulin
Changes in body fat distribution | 8 weeks
  Abdominal axial T1-weighted slices

CONTACTS AND LOCATIONS:
Locations (1):
- Quebec Heart and Lung Institute - Laval University, Québec, Canada

IPD SHARING:
Plan to Share IPD: No